CLINICAL TRIAL: NCT03836222
Title: A Phase I, Single Centre, Open-Label, Non-Randomised Study to Evaluate the PK of Single and Optional Multiple Dosing Regimens of MR Formulations of PCS499 Compared to Trental® (Pentoxifylline) Administered to Healthy Subjects Under Fed Conditions
Brief Title: Study to Evaluate the PK of Single and Optional Multiple Dosing Regimens of MR Formulations of PCS499 Compared to Trental® Administered to Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Processa Pharmaceuticals (Industry)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: PCS499.1005
Record Dates: First submitted 2019-01-31; First posted 2019-02-11 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Healthy
MeSH Terms: interventions — Pentoxifylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- PCS499 MR Tablet Prototype 2 (Experimental): 600 mg single dose
  Interventions: Drug: PCS499
- Trental MR tablet 400mg (Active Comparator): single dose
  Interventions: Drug: Trental
- PCS499 MR Tablet Prototype 4 (Experimental): 600mg single dose
  Interventions: Drug: PCS499
- PCS499 MR Tablet Prototype 1 (Experimental): 600mg single dose
  Interventions: Drug: PCS499
- Trental MR Tablet (Active Comparator): 400 mg multiple dose
  Interventions: Drug: Trental
- PCS499 MR Tablet 900mg (Experimental): multiple dose
  Interventions: Drug: PCS499
- PCS499 MR Tablet 600mg (Experimental): multiple dose
  Interventions: Drug: PCS499

INTERVENTIONS:
Drug: PCS499 — MR tablet
  Arms: PCS499 MR Tablet 600mg; PCS499 MR Tablet 900mg; PCS499 MR Tablet Prototype 1; PCS499 MR Tablet Prototype 2; PCS499 MR Tablet Prototype 4
Drug: Trental — comparator tablet
  Arms: Trental MR Tablet; Trental MR tablet 400mg

SUMMARY:
This was a Phase I, single centre, open-label, non-randomised study and was designed to be conducted in up to 2 parts. The purpose of Part 1 was to identify a MR formulation of PCS499 that would provide an optimal dosing regimen in patients. The purpose of Part 2 of the study was to generate repeat dose information for the selected MR formulation of PCS499 in order to provide additional PK information for future patient studies.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant, non-lactating female subjects
2. Aged 18 to 55 years, inclusive
3. Subjects who were healthy as determined by no clinically relevant abnormalities identified by a detailed medical history, full physical examination, vital signs, 12-lead resting electrocardiogram (ECG; corrected QT interval [QTc] ≤450, QRS <120, PR <220; normal morphology) performed at the screening visit and prior to each dosing
4. Body mass index (BMI) of 18.0 to 35.0 kg/m2 inclusive or, if outside the range, considered not clinically significant by the investigator and body weight >50 kg
5. Subjects who were willing and able to be confined at the clinical research centre for the scheduled inpatient visits
6. Ability to swallow multiple tablets whole

Exclusion Criteria:

1. Subject had a clinically significant history of GI, cardiovascular, musculoskeletal, endocrine, hematologic, psychiatric, renal, hepatic, bronchopulmonary, neurologic, immunologic, and/or lipid metabolism disorders and/or drug hypersensitivity
2. Subject had a known or suspected malignancy with the exception of basal cell carcinoma
3. Subject had a positive blood screen for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus antibody (HCV Ab) at the screening visit
4. Female subjects who were pregnant or lactating (all female subjects required a negative serum pregnancy test at the screening and a negative urine pregnancy test at each admission).
5. Subject had active disease or symptoms within 7 days prior to Day -1, such as nausea, vomiting, diarrhoea, and infection
6. Subject had undergone a hospital admission or major surgery within 30 days prior to the Screening visit
7. Subjects who had taken part in Part 1 were not permitted to take part in Part 2

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2018-06-04 (Actual); Study Completion 2018-06-04 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentrations (Cmax) for Part 1 | Blood samples will be drawn prior to single dose administration of study drug and at 11 other timepoints in a 24 hour period.
  Serial blood sampling at specified time points for determination of plasma concentration-time profiles
Maximum plasma concentrations (Cmax) in Part 2 | Blood sampling will be drawn prior to the single dose administration on Days 1 & 4 and at 11 other timepoints in the following 24 hours. In addition, pre-dose trough samples will be taken on Days 2 &3.
  Serial blood sampling at specified time points for determination of plasma concentration-time profiles

CONTACTS AND LOCATIONS:
Overall Officials: Sharan Sidhu, MBChB, Principal Investigator — Quotient Sciences
Locations (1):
- Quotient Sciences, Ruddington, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No